CLINICAL TRIAL: NCT04413370
Title: The Development of Artificial Intelligence Dry Eye Screening and Referral System
Brief Title: Dry Eye Screening and Referral System
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Professor, Sun Yat-sen University
Other Study IDs: Dry eye screening system
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe Group: This group of subjects needed a referral to the hospital for further treatments.
  Interventions: Diagnostic Test: Dry eye diagnostic test
- Mild group: This group of subjects was diagnosed with dry eye but can use artificial tears instead of further treatment.
  Interventions: Diagnostic Test: Dry eye diagnostic test
- Follow-up group: This group of subjects had no dry eye symptoms and signs and belonged to the normal control group.
  Interventions: Diagnostic Test: Dry eye diagnostic test

INTERVENTIONS:
Diagnostic Test: Dry eye diagnostic test — The artificial intelligent dry eye screening platform

SUMMARY:
Dry eye is one of the most common ocular surface diseases. Its pathogenic factors are related to multiple etiology. Because of the complexity of the pathogenesis of dry eye, the diversity of related examinations, and the inconsistency of symptoms and signs of dry eye patients, the diagnosis of dry eye has higher requirements on the professional technology and examination equipment of ophthalmologists.

The purpose of this study is to establish a case-control cohort of dry eye patients. Multimodal data will be collected from participants, including medical history information, ocular surface disease index scale (OSDI), anterior segment photography, and treatment outcome of dry eye patients. The correlation between the characteristics of anterior segment images and dry eye diagnosis will be explored by artificial intelligence algorithms. The purpose of this study was to develop an artificial intelligence dry eye screening and referral system.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects whose age are greater than or equal to 18 years old;
2. Subjects who can cooperate with the inspection;
3. Subjects who agree to participate in the study and sign the consent form.

Exclusion Criteria:

1. Subjects who cannot do the inspection.
2. Subjects who suffer from diseases that compromise the inspection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who are equal or over 18 years old with or without dry eye symptoms and signs.
Sampling Method: Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (severe) | up to 1 month
  AUC values for predicting whether subject need to be referral or not.

SECONDARY OUTCOMES:
Area under the curve (each group) | up to 1 month
  AUC values for predicting whether subject can be accurately grouped into each of the four groups.
Accuracy, true positive rate, and true negative rate | up to 1 month
  The performance of this artificial platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No